CLINICAL TRIAL: NCT07364773
Title: Enhancing Rehabilitation Participation in Patients With Spinal Cord Injury or Disorder Using Motivational Interviewing
Brief Title: Enhancing Rehabilitation Participation in Patients With SCI/D Using Motivational Interviewing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Baylor Research Institute (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Linda Ehrlich-Jones, PhD, Associate Director, Center for Rehabilitation Outcomes Research, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STU00219326; 973467 (Other Grant/Funding Number: Craig H. Neilsen Foundation)
Record Dates: First submitted 2025-10-09; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injuries (SCI); Spinal Cord Disease
Keywords: Spinal Cord Injury; Spinal Cord Disorder; Motivational Interviewing; Rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Patients in the experimental group will receive treatment from a Physical or Occupational Therapist trained in Motivational Interviewing. Those in the control group will receive standard therapy communication.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient participants and the assessor rating participation level during therapy sessions will be blinded. Therapist participants will be aware of the arm in which they will be placed through training on motivational interviewing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: Motivational Interviewing (Experimental): Physical and Occupational Therapists in this group will receive 16 hours of training in Motivational Interviewing and use these techniques during sessions with enrolled patient participants.
  Interventions: Behavioral: Motivational Interviewing
- Control Group: Standard Care (No Intervention): Therapists in this group will not participate in additional training and provide standard care to enrolled patient participants.

INTERVENTIONS:
Behavioral: Motivational Interviewing — Motivational Interviewing is an evidence-based counseling style that aims to foster positive health behavior change in patients through their desires and actions.
  Arms: Experimental Group: Motivational Interviewing

SUMMARY:
The purpose of this multi-site clinical trial is to see whether people with spinal cord injury or disorder (SCI/D) demonstrate higher level of participation in rehabilitation sessions and other outcomes when their therapists are trained in a counseling style called motivational interviewing. We want to answer the following questions:

1. Do inpatients with SCI/D treated by physical therapists (PTs) and occupational therapists (OTs) who receive MI training and coaching demonstrate greater therapy participation compared to those treated by therapists who do not receive MI training and coaching?
2. Do inpatients with SCI/D treated by PTs and OTs who receive MI training and coaching demonstrate greater functional improvement at discharge from inpatient rehabilitation and greater community integration at 6 months after discharge compared to those treated by therapists who do not receive MI training and coaching?
3. What are the potential moderators and mediators of the effect of training and coaching on MI skills on therapy participation?

Researchers will compare patient participation level and other outcomes of inpatients with SCI/D treated by PTs and OTs who receive MI training and coaching with those treated by therapists who do not receive MI training and coaching.

Therapist participants will:

1. Audio record 2 therapy sessions per week with each enrolled SCI patient participant
2. Half of the therapists will attend a 16-hour training on MI skills and 2 practice therapy session

Patient participants will:

1. Consent to audio recording of their therapy sessions
2. Complete one brief survey near the time of their discharge and another survey 6 months later

DETAILED DESCRIPTION:
We plan to conduct a multi-site randomized controlled trial of motivational interviewing (MI) training for physical therapists (PTs) and occupational therapists (OTs) who treat people with SCI during inpatient rehabilitation. We will test whether patients treated by MI trained PTs and OTs demonstrate greater participation in therapy sessions and better functional, social, and educational/occupational outcomes relative to patients treated by therapists without MI training. This stage of research is appropriate because a Neilsen Foundation funded pilot study that we recently completed had promising results. Study results showed that SCI patients treated by MI trained PTs and OTs participated significantly more actively in therapy sessions compared to controls. However, the study had several limitations that need to be addressed to produce a more definitive and influential trial. First, the study was conducted at a single site and results may not generalize to other sites. Second, we did not examine whether MI training and improved participation resulted in patients having better clinically meaningful outcomes such as higher likelihood of discharge to home or superior functional, social, or educational/occupational outcomes. Third, therapists trained in MI achieved only minimal competency in MI skills. We hypothesize that if therapists received ongoing coaching to improve their MI skills during the trial the positive impact on patient participation and other outcomes might be even more robust.

ELIGIBILITY:
Therapist Inclusion Criteria:

* Inpatient therapist specializing in spinal cord injury patients for at least 3 months;
* Practicing at the designated SCI inpatient units at Shirley Ryan AbilityLab, Baylor Scott & White Institute for Rehabilitation and University of Washington-Harborview Medical Center;
* Willing to audio record conversations during regularly-scheduled rehabilitation therapy sessions with patients;
* Willing and able to participate in 16 hours of MI training; and
* Willing to receive feedback on MI skills.

Therapist Exclusion Criteria:

* Inability to speak and understand English
* Inpatient therapist specializing in spinal cord injury patients for less than 3 months; and
* Unwilling or unable to follow the study protocol

Patient Inclusion Criteria:

* Adults (18+)
* Presence of a traumatic or non-traumatic spinal cord injury
* Inpatient in the spinal cord injury unit of the three study sites
* Has a physical or occupational therapist who is a participant in the study

Patient Exclusion Criteria:

* Inability to speak and understand English
* Cognitive deficits
* Unwilling to allow for therapy sessions to be recorded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-04-20 (Estimated); Study Completion 2027-04-20 (Estimated)

PRIMARY OUTCOMES:
Therapy Participation Level | From enrollment to the end of 4-week treatment
  A blinded assessor will use the Pittsburgh Rehabilitation Participation Scale (PRPS) to measure therapy participation in inpatients with SCI treated by therapists trained in Motivational Interviewing (MI) compared to those treated by therapists not trained to use MI. The PRPS rating ranges from 1 (none) to 6 (excellent), with higher scores indicating higher level of participation

SECONDARY OUTCOMES:
Efficacy of Motivational Interviewing (MI) Training | During 1 year of inpatient rehabilitation
  We will use the Motivational Interviewing Treatment Integrity (MITI) to continually evaluate the efficacy of MI training by measuring adherence to MI counseling skills in rehabilitation therapists trained to use MI compared to those not trained to use MI. The ratings are on a 5-point Likert scale from 1 (low) to 5 (high), with higher scores indicating higher level of efficacy.
Functional Abilities | At week 4
  The Spinal Cord Injury Functional Independence (SCI-FI) will be administered to patient participants within approximately one week of their discharge from inpatient rehabilitation. The response scale range from 1 (unable to do the activity) to 5 (no difficulty), with higher scores indicating higher functional ability.
Participation in the Community | At 6 months post-discharge
  The Participation Assessment with Recombined Tools-Objective (PART-O) will be administered to patient participants to measure their level of involvement in the community 6 months post discharge. Higher scores indicate higher level of participation.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Ehrlich-Jones, PhD, RN, Principal Investigator — Shirley Ryan AbilityLab
Locations (3):
- United States (3):
  - Shirley Ryan AbilityLab, Chicago, Illinois
  - Baylor Scott & White Institute for Rehabilitation, Dallas, Texas
  - University of Washington - Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moyers TB, Rowell LN, Manuel JK, Ernst D, Houck JM. The Motivational Interviewing Treatment Integrity Code (MITI 4): Rationale, Preliminary Reliability and Validity. J Subst Abuse Treat. 2016 Jun;65:36-42. doi: 10.1016/j.jsat.2016.01.001. Epub 2016 Jan 13. PMID 26874558
- [Background] Ryan RM, Deci EL. Self-determination theory and the facilitation of intrinsic motivation, social development, and well-being. Am Psychol. 2000 Jan;55(1):68-78. doi: 10.1037//0003-066x.55.1.68. PMID 11392867
- [Background] Deci EL, Ryan RM. Self-determination theory in health care and its relations to motivational interviewing: a few comments. Int J Behav Nutr Phys Act. 2012 Mar 2;9:24. doi: 10.1186/1479-5868-9-24. PMID 22385839
- [Background] Miller WR, Rollnick S. Motivational Interviewing: Helping People Change. Third ed. New York, NY: The Guilford Press; 2013.
- [Background] Miller WR, Rollnick S. Meeting in the middle: motivational interviewing and self-determination theory. Int J Behav Nutr Phys Act. 2012 Mar 2;9:25. doi: 10.1186/1479-5868-9-25. No abstract available. PMID 22385872
- [Background] Kramer Schmidt L, Andersen K, Nielsen AS, Moyers TB. Lessons learned from measuring fidelity with the Motivational Interviewing Treatment Integrity code (MITI 4). J Subst Abuse Treat. 2019 Feb;97:59-67. doi: 10.1016/j.jsat.2018.11.004. Epub 2018 Nov 20. PMID 30577900
- [Background] Whiteneck GG, Gassaway J, Ketchum JM. Transforming a Traumatic Brain Injury Measure of Participation Into a Psychometrically Sound Spinal Cord Injury Participation Measure. Arch Phys Med Rehabil. 2019 Dec;100(12):2293-2300. doi: 10.1016/j.apmr.2019.06.020. Epub 2019 Aug 14. PMID 31421095
- [Background] Heinemann AW, Dijkers MP, Ni P, Tulsky DS, Jette A. Measurement properties of the Spinal Cord Injury-Functional Index (SCI-FI) short forms. Arch Phys Med Rehabil. 2014 Jul;95(7):1289-1297.e5. doi: 10.1016/j.apmr.2014.01.031. Epub 2014 Mar 3. PMID 24602551
- [Background] Miller WR, Yahne CE, Moyers TB, Martinez J, Pirritano M. A randomized trial of methods to help clinicians learn motivational interviewing. J Consult Clin Psychol. 2004 Dec;72(6):1050-62. doi: 10.1037/0022-006X.72.6.1050. PMID 15612851
- [Background] Bombardier CH, Dyer JR, Burns P, Crane DA, Takahashi MM, Barber J, Nash MS. A tele-health intervention to increase physical fitness in people with spinal cord injury and cardiometabolic disease or risk factors: a pilot randomized controlled trial. Spinal Cord. 2021 Jan;59(1):63-73. doi: 10.1038/s41393-020-0523-6. Epub 2020 Jul 21. PMID 32694748
- [Background] Bombardier CH, Bell KR, Temkin NR, Fann JR, Hoffman J, Dikmen S. The efficacy of a scheduled telephone intervention for ameliorating depressive symptoms during the first year after traumatic brain injury. J Head Trauma Rehabil. 2009 Jul-Aug;24(4):230-8. doi: 10.1097/HTR.0b013e3181ad65f0. PMID 19625862
- [Background] O'Halloran PD, Blackstock F, Shields N, Holland A, Iles R, Kingsley M, Bernhardt J, Lannin N, Morris ME, Taylor NF. Motivational interviewing to increase physical activity in people with chronic health conditions: a systematic review and meta-analysis. Clin Rehabil. 2014 Dec;28(12):1159-71. doi: 10.1177/0269215514536210. Epub 2014 Jun 18. PMID 24942478
- [Background] Ehrlich-Jones L, Mallinson T, Fischer H, Bateman J, Semanik PA, Spring B, Ruderman E, Chang RW. Increasing physical activity in patients with arthritis: a tailored health promotion program. Chronic Illn. 2010 Dec;6(4):272-81. doi: 10.1177/1742395309351243. Epub 2010 Aug 9. PMID 20696695
- [Background] Watkins CL, Auton MF, Deans CF, Dickinson HA, Jack CI, Lightbody CE, Sutton CJ, van den Broek MD, Leathley MJ. Motivational interviewing early after acute stroke: a randomized, controlled trial. Stroke. 2007 Mar;38(3):1004-9. doi: 10.1161/01.STR.0000258114.28006.d7. Epub 2007 Feb 15. PMID 17303766
- [Background] Bombardier CH, Rimmele CT. Alcohol use and readiness to change after spinal cord injury. Arch Phys Med Rehabil. 1998 Sep;79(9):1110-5. doi: 10.1016/s0003-9993(98)90180-0. PMID 9749693
- [Background] Bombardier CH, Ehde DM, Gibbons LE, Wadhwani R, Sullivan MD, Rosenberg DE, Kraft GH. Telephone-based physical activity counseling for major depression in people with multiple sclerosis. J Consult Clin Psychol. 2013 Feb;81(1):89-99. doi: 10.1037/a0031242. PMID 23379265
- [Background] Soderlund LL, Madson MB, Rubak S, Nilsen P. A systematic review of motivational interviewing training for general health care practitioners. Patient Educ Couns. 2011 Jul;84(1):16-26. doi: 10.1016/j.pec.2010.06.025. Epub 2010 Jul 25. PMID 20667432
- [Background] Schwarzer R, Lippke S, Luszczynska A. Mechanisms of health behavior change in persons with chronic illness or disability: the Health Action Process Approach (HAPA). Rehabil Psychol. 2011 Aug;56(3):161-70. doi: 10.1037/a0024509. PMID 21767036
- [Background] Lequerica AH, Kortte K. Therapeutic engagement: a proposed model of engagement in medical rehabilitation. Am J Phys Med Rehabil. 2010 May;89(5):415-22. doi: 10.1097/PHM.0b013e3181d8ceb2. PMID 20407308
- [Background] Teeter L, Gassaway J, Taylor S, LaBarbera J, McDowell S, Backus D, Zanca JM, Natale A, Cabrera J, Smout RJ, Kreider SE, Whiteneck G. Relationship of physical therapy inpatient rehabilitation interventions and patient characteristics to outcomes following spinal cord injury: the SCIRehab project. J Spinal Cord Med. 2012 Nov;35(6):503-26. doi: 10.1179/2045772312Y.0000000058. PMID 23318034
- [Background] Ozelie R, Gassaway J, Buchman E, Thimmaiah D, Heisler L, Cantoni K, Foy T, Hsieh CH, Smout RJ, Kreider SE, Whiteneck G. Relationship of occupational therapy inpatient rehabilitation interventions and patient characteristics to outcomes following spinal cord injury: the SCIRehab project. J Spinal Cord Med. 2012 Nov;35(6):527-46. doi: 10.1179/2045772312Y.0000000062. PMID 23318035
- [Background] Granger CV, Karmarkar AM, Graham JE, Deutsch A, Niewczyk P, Divita MA, Ottenbacher KJ. The uniform data system for medical rehabilitation: report of patients with traumatic spinal cord injury discharged from rehabilitation programs in 2002-2010. Am J Phys Med Rehabil. 2012 Apr;91(4):289-99. doi: 10.1097/PHM.0b013e31824ad2fd. PMID 22407160
- [Background] Seel RT, Corrigan JD, Dijkers MP, Barrett RS, Bogner J, Smout RJ, Garmoe W, Horn SD. Patient Effort in Traumatic Brain Injury Inpatient Rehabilitation: Course and Associations With Age, Brain Injury Severity, and Time Postinjury. Arch Phys Med Rehabil. 2015 Aug;96(8 Suppl):S235-44. doi: 10.1016/j.apmr.2014.10.027. PMID 26212400
- [Background] Lenze EJ, Munin MC, Quear T, Dew MA, Rogers JC, Begley AE, Reynolds CF 3rd. The Pittsburgh Rehabilitation Participation Scale: reliability and validity of a clinician-rated measure of participation in acute rehabilitation. Arch Phys Med Rehabil. 2004 Mar;85(3):380-4. doi: 10.1016/j.apmr.2003.06.001. PMID 15031821
- [Background] Lequerica AH, Rappor LJ, Whitman R. Psychometric properties of the Rehabilitation Therapy Engagement Scale among patients with acquired brain injury. Rehabil Psychol. 2007;51:331-337.
- [Background] Kortte KB, Falk LD, Castillo RC, Johnson-Greene D, Wegener ST. The Hopkins Rehabilitation Engagement Rating Scale: development and psychometric properties. Arch Phys Med Rehabil. 2007 Jul;88(7):877-84. doi: 10.1016/j.apmr.2007.03.030. PMID 17601468

DOCUMENTS (3):
  • Study Protocol (2024-12-12): https://cdn.clinicaltrials.gov/large-docs/73/NCT07364773/Prot_000.pdf
  • Informed Consent Form: Consent Form for Therapist Participant (2024-12-12): https://cdn.clinicaltrials.gov/large-docs/73/NCT07364773/ICF_001.pdf
  • Informed Consent Form: Consent Form for Patient Participant (2024-12-12): https://cdn.clinicaltrials.gov/large-docs/73/NCT07364773/ICF_002.pdf